CLINICAL TRIAL: NCT00533052
Title: Addressing Emotional and Cognitive Factors in Behavioral Weight Loss Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23 DK73536 (completed); K23DK073536 (NIH)
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Overweight; Obesity
Keywords: Behavioral weight loss
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Affective and Cognitive Skills Training (Experimental): Standard Behavioral Weight Loss Treatment Plus Affective and Cognitive Skills Training
  Interventions: Behavioral: Affective and Cognitive Skills Training

INTERVENTIONS:
Behavioral: Affective and Cognitive Skills Training — 24-week, weekly, group behavioral weight loss treatment with affective and cognitive skills training

SUMMARY:
Behavioral weight loss, the current treatment of choice for moderate obesity, achieves impressive short term results, however, weight regain following treatment is a major problem. Over 50% of participants in behavioral weight loss programs report difficulty with internal antecedents to unhealthy weight control behaviors and this difficulty is associated with weight regain following treatment. Current treatment approaches do not adequately address these antecedents. The aim of this series of studies is to develop, implement, and evaluate a behavioral weight loss program modified to provide participants with skills to deal effectively with affective and cognitive difficulties. The study targets men and women with BMI of 27-40 who self-report difficulty with emotional and/or cognitive antecedents to unhealthy weight control behaviors. The study is an uncontrolled pilot study in 20 participants to initially assess acceptability and efficacy of the innovative treatment. The long-term goal of this research is to improve the weight loss maintenance outcomes of behavioral weight loss programs by addressing affective and cognitive antecedents to unhealthy weight control behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 70 years
* Body mass index between 27 and 40
* Score 5 or above on the internal disinhibition scale of the Eating Inventory

Exclusion Criteria:

* Are currently participating in a weight loss program and/or are taking a weight loss medication or lost greater than or equal to 5% of body weight during the past six months
* Are pregnant, lactating, less than 6 months postpartum or plan to become pregnant during the time frame of the investigation
* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q). Individuals endorsing joint problems, prescription medication usage, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 6 months

SECONDARY OUTCOMES:
Internal disinhibition as measured by the Eating Inventory | 6 months
  The internal disinhibition subscale of the Eating Inventory ranges from 0 to 8, with high values indicating more disinhibition.
Treatment acceptability based on qualitative feedback | 6 months
Attendance data | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Heather M. Niemeier, Ph.D., Principal Investigator — The Miriam Hospital/The Warren Alpert Medical School of Brown University
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Niemeier HM, Leahey T, Palm Reed K, Brown RA, Wing RR. An acceptance-based behavioral intervention for weight loss: a pilot study. Behav Ther. 2012 Jun;43(2):427-35. doi: 10.1016/j.beth.2011.10.005. Epub 2011 Dec 1. PMID 22440077